CLINICAL TRIAL: NCT02546245
Title: Modification and Evaluation of the Educational Mobile Games Heroes of Knowledge in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1503015556
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Math Knowledge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heroes of Knowledge Game (Experimental)
  Interventions: Behavioral: Heroes of Knowledge
- Attention/Time Control Games (Active Comparator)
  Interventions: Behavioral: Attention/Time Control Game

INTERVENTIONS:
Behavioral: Heroes of Knowledge — Participants will play their assigned game(s) on a tablet computer for 1-1.5 hours, 2-3 times per week for 2-4 weeks (to accumulate 6-8 hours of gameplay).
  Arms: Heroes of Knowledge Game
Behavioral: Attention/Time Control Game — Participants will play their assigned game(s) on a tablet computer for 1-1.5 hours, 2-3 times per week for 2-4 weeks (to accumulate 6-8 hours of gameplay).
  Arms: Attention/Time Control Games

SUMMARY:
The goal of the proposed research is to adapt and rigorously evaluate educational mobile games, designed as a downloadable mobile apps to be played on smartphones or tablets. Investigators will be partnering with Yogome for this project. Yogame is a company dedicated to creating educational games that aim to reinforce knowledge acquired in school and help children learn new things in an entertaining and fun way.

DETAILED DESCRIPTION:
This study will modify and evaluate the Heroes of Knowledge (HoK) games, beginning with the Math Heroes game which was designed to be played for up to 8 hours. Other games in the HoK series may be included in this process if they are fully developed and available for testing. In testing the efficacy of the Math Heroes game, children will play the game for 1-1.5 hours per week, 2-3 times per week, for 2-4 weeks (to accumulate 6-8 hours of game play). The game has been designed to target math knowledge skills identified by the Common Core Standards for Mathematics (2012).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in first grade and interested and able to participate in a mobile app-based videogame (willing to sit with a tablet computer for approximately 1-1.5 hours, 2-3 times per week for 2-4 weeks).

Exclusion Criteria:

* None

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pearson KeyMath3 Diagnostic Assessment (KeyMath-3DA) | Baseline
  A comprehensive, norm-referenced measure of essential mathematical concepts and skills. Test items are grouped into 10 subtests that represent three general math content areas: Basic Concepts (conceptual knowledge), Operations (computational skills), and Applications (problem solving).
Pearson KeyMath3 Diagnostic Assessment (KeyMath-3DA) | 2-4 weeks
  A comprehensive, norm-referenced measure of essential mathematical concepts and skills. Test items are grouped into 10 subtests that represent three general math content areas: Basic Concepts (conceptual knowledge), Operations (computational skills), and Applications (problem solving).

SECONDARY OUTCOMES:
Academic Self Competence will be captured using a "structure alternate format" scale | Baseline
  Self-Competence will be captured using a "structure alternate format" scale designed for young children adapted from the 28-item Perceived Competence Scale in Children. For this study, self-competence is defined as a child's sense of cognitive competence. Each item is scored from 1 to 4, where a score of 1 indicates low perceived competence and a score of 4 reflects high perceived competence. Scores are summed and then averaged.
Academic Self Competence will be captured using a "structure alternate format" scale | 2-4 weeks
  Self-Competence will be captured using a "structure alternate format" scale designed for young children adapted from the 28-item Perceived Competence Scale in Children. For this study, self-competence is defined as a child's sense of cognitive competence. Each item is scored from 1 to 4, where a score of 1 indicates low perceived competence and a score of 4 reflects high perceived competence. Scores are summed and then averaged.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Fiellin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States